CLINICAL TRIAL: NCT02575417
Title: Development of a Community Engagement Activity for Advance Care Planning
Acronym: CERC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Lauren Van Scoy, Assistant Professor, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00003004
Record Dates: First submitted 2015-10-12; First posted 2015-10-14 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Chronic Disease
Keywords: advance care planning; end-of-life care; health games; Family caregivers; Advance directives
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Patient Only (Experimental): Individuals who meet the following criteria will play "My Gift of Grace," a conversation game.
  Eligibility Criteria for Patient Only Groups:
  1. are 18 years or older
  2. speak and read English
  3. have at least one chronic illness (cancer, chronic pulmonary disease, coronary artery disease, congestive heart failure, peripheral vascular disease, severe chronic liver disease, diabetes with end organ damage, renal failure)
  4. have not completed an advance directive within the past 18 months
  5. are able to sit for about 2.5-3 hours
  6. are able to focus on the game for about 1.5-2 hours
  7. can complete required surveys
  Interventions: Behavioral: Conversation Game
- Caregiver Only (Experimental): Individuals who meet the following criteria will play "My Gift of Grace," a conversation game.
  Eligibility Criteria for Caregiver Only Groups:
  1. are 18 years or older
  2. speak and read English
  3. have been an unpaid caregiver for an adult over the age of 18 in the last 12 months. Being an unpaid caregiver may include helping with personal needs or household chores, managing a person's finances, arranging for outside services, or visiting regularly to see how they are doing. This person need not live with participants in order for them to identify as caregivers;
  4. are able to sit for about 2.5-3 hours
  5. are able to focus on the game for about 1.5-2 hours
  6. can complete required survey
  7. care recipient is capable of discussing medical issues
  8. care recipient has not completed an AD in past 18 months
  Interventions: Behavioral: Conversation Game
- Surrogate Decision Maker with Patient (Experimental): Individuals who meet the following criteria will play "My Gift of Grace," a conversation game.
  Eligibility Criteria for Surrogate Decision Maker and Patient Group:
  1. considers themselves a surrogate decision maker for an adult with a chronic illness (defined in "Patient Only" Group)
  2. are 18 years or older
  3. speak and read English
  4. are able to sit for about 2.5-3 hours
  5. are able to focus on the game for about 1.5-2 hours
  6. can complete required surveys
  7. both patient and surrogate decision maker are able to attend study session together
  8. patient must meet eligibility criteria defined in "Patient Only" group
  Interventions: Behavioral: Conversation Game

INTERVENTIONS:
Behavioral: Conversation Game — The game consists of 47 question cards that prompt players to identify and articulate their values and beliefs related to dying and end-of-life issues; 20 questions have been selected for this study

SUMMARY:
This study will determine the feasibility of using an end-of-life conversation game (called "My Gift of Grace") as a community engagement activity series to help caregivers, patients with chronic illness, and/or their families perform advance care planning.

DETAILED DESCRIPTION:
While many patients and caregivers of individuals with chronic illness recognize the importance of advance care planning, many feel uncomfortable initiating end-of-life conversations with loved ones. Few tools exist that effectively engage caregivers and address their particular concerns and needs. The investigators have preliminary data showing that an easily implementable intervention (a conversation game) effectively engages healthy participants in realistic and satisfying ACP conversations. However, the investigators have not yet tested the acceptability or feasibility of using the game in a population of caregivers and/or patients with chronic illness. This pilot project will enable us to engage community-based patients and caregivers to determine if they find the game a satisfying, acceptable, relevant, and effective tool for advance care planning.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to participate if they fall into at least one of the following three groups:

1. CAREGIVER criteria include:

   1. are 18 years or older
   2. speak and read English
   3. have been an unpaid caregiver for an adult over the age of 18 in the last 12 months. Being an unpaid caregiver may include helping with personal needs or household chores, managing a person's finances, arranging for outside services, or visiting regularly to see how they are doing. This person need not live with participants in order for them to identify as caregivers;
   4. are able to sit for about 2.5-3 hours
   5. are able to focus on the game for about 1.5-2 hours
   6. can complete required survey
   7. care recipient is capable of discussing medical issues
   8. care recipient has not completed an AD in past 18 months
2. PATIENT criteria include:

   1. are 18 years or older
   2. speak and read English
   3. have at least one chronic illness (cancer, chronic pulmonary disease, coronary artery disease, congestive heart failure, peripheral vascular disease, severe chronic liver disease, diabetes with end organ damage, renal failure-defined using Iezonnis' ICD-9 criteria67)
   4. have not completed an advance directive within the past 18 months
   5. are able to sit for about 2.5-3 hours
   6. are able to focus on the game for about 1.5-2 hours
   7. can complete required surveys
3. SURROGATE DECISION MAKERS FOR PATIENTS WITH CHRONIC ILLNESS criteria include:

   1. considers themselves a surrogate decision maker for an adult with a chronic illness (defined above)
   2. are 18 years or older
   3. speak and read English
   4. are able to sit for about 2.5-3 hours
   5. are able to focus on the game for about 1.5-2 hours
   6. can complete required surveys

Exclusion Criteria:

1. Do not fall into any of the three categories above
2. Have a diagnosis of dementia (by self-report or chart review)
3. Fall into the Surrogate Decision Maker category but the patient cannot also participate in the same study session

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in self-efficacy and readiness to perform advance care planning behaviors | Baseline (before study session) and 12 weeks post-study
  55-item survey, likert scale ratings

SECONDARY OUTCOMES:
Experiences and perceptions of intervention | 10 minutes after intervention ends
  Focus-group, open-ended qualitative questions

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Van Scoy, MD, Principal Investigator — Penn State Hershey College of Medicine
Locations (1):
- Penn State Hershey College of Medicine, Hershey, Pennsylvania, United States

REFERENCES:
- [Result] Van Scoy LJ, Reading JM, Hopkins M, Smith B, Dillon J, Green MJ, Levi BH. Community Game Day: Using an End-of-Life Conversation Game to Encourage Advance Care Planning. J Pain Symptom Manage. 2017 Nov;54(5):680-691. doi: 10.1016/j.jpainsymman.2017.07.034. Epub 2017 Jul 23. PMID 28743662